CLINICAL TRIAL: NCT01142557
Title: Therapy of the Chronic Multiple Sclerosis With Interferon-beta 1a (Rebif®)
Brief Title: An Observational Study to Document the Effectiveness and Compatibility of Rebif 44 or 22 µg in the Therapy of the Chronic Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Gesellschaft für Therapieforschung mbH (Industry)
Responsible Party: Dr. Norbert Zessack/Head of Medicine BU Neurology, Merck Serono GmbH Germany, an affiliate of MerckKGaA, Darmstadt, Germany
Other Study IDs: REBIJECT II
Record Dates: First submitted 2010-06-10; First posted 2010-06-11 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2010-06

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Rebif; Interferon-beta
MeSH Terms: conditions — Multiple Sclerosis | interventions — Interferon beta-1a

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Drug: Interferon beta-1a (Rebif) — A dosage of 44 µg or 22 µg interferon beta-1a (Rebif) as subcutaneous self-injection three times a week was recommended for therapy of the included, suitable MS subjects after a creep-in phase of 4 weeks.
  Other Names: Rebif

SUMMARY:
The aim of this case series was to document the effectiveness and compatibility of Rebif 44 or 22 µg in the therapy of the chronic multiple sclerosis (MS) under practical conditions on a large collection of subjects. In addition, the side effects possibly occurring in the initial phase of therapy and satisfaction of the subject as well as the treating doctor was also documented.

DETAILED DESCRIPTION:
Interferon beta-1a is established as therapy of the first choice in the treatment of the chronic MS. The PRISMS study has shown that the therapy with Rebif reduces the frequency and seriousness of clinical attacks or episodes over 4 years and the progress of the disability slows down. This clinically identifiable effectiveness is supported by the significant decrease in the nuclear spin-tomographically provable disease activity and total lesion stress. The interferon-beta therapy cannot heal the MS but the therapy with Rebif can however reduce number and seriousness of attacks or episodes and can clearly delay progress of the disability. The Rebif therapy is a long-term treatment, as a result the subject may not feel the positive effects immediately, but effects of the therapy can only be noticed after a longer period.

At the beginning of the therapy, interferon-beta-specific side effects such as fever, fever-like symptoms, muscle and joint pains as well as reactions at the injection points can occur. The described reactions are individually dependent on respective subjects in duration and seriousness, however they are normally mild and temporary.

OBJECTIVE

The objective of this study was to document the effectiveness and compatibility of Rebif 44 or 22 µg proven in clinical studies in the therapy of the chronic MS under practical conditions on a large collection of subjects. Especially the handling of injection aid of Rebiject II when using with Rebif pre-filled syringe was documented.

The observation period in this study was 3 months per subject and approximately 500 subjects with clinically safe diagnosis of a chronic MS and ability to walk (also with aids) were recorded in the case series. Demographic data as well as details about the diagnosis, course, current status and previous therapy of MS was recorded at the beginning of the case series. All data collected within the framework of the therapy, such as e.g. of blood count test or determination of the liver function test values for checking the possible influence of Rebif on these parameters was part of the case series and hence were documented.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with clinically safe diagnosis of a chronic MS and ability to walk (also with aids).

Exclusion Criteria:

* Subjects with primary chronically progressive course of the MS
* Pregnant or nursing female subjects
* Subjects with severe depressions
* Epilepsy subjects whose symptoms cannot be cured adequately with therapy
* Subjects with existing systemic concurrent diseases (e.g. diabetes, heart, liver, kidney diseases)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with clinically safe diagnosis of a chronic MS and ability to walk were recorded in the case series.
Sampling Method: Probability Sample
Enrollment: 522 (Actual)
Dates: Start 2004-06; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Assessment of the effectiveness and compatibility of Rebif 44 or 22 µg | Baseline to 3 months

SECONDARY OUTCOMES:
Side effects occurring in the initial phase of therapy | Baseline to 3 months
Satisfaction of the subject as well as the treating doctor | Baseline to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Zessack, Study Director — Merck Serono GmbH, Germany
Locations (1):
- Merck Serono GmbH, Darmstadt, Germany